CLINICAL TRIAL: NCT06064955
Title: Pair 2 Care: Peer Support for Caregivers of Black Americans Living With Dementia
Acronym: Pair 2 Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Cambia Health Foundation (Other)
Responsible Party: Principal Investigator, Karen Moss, Assistant Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023B0071
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Family Caregiver; Dementia; Peer Support
Keywords: African American/Black
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: A model to explain factors impacting advance care planning among African Americans
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer Support (Experimental): Former caregivers will be paired with a current caregivers
  Interventions: Behavioral: Peer Support

INTERVENTIONS:
Behavioral: Peer Support — Former caregivers will be paired with a current caregiver based on a similar personal attribute (e.g., relationship to care recipient). Each pair will complete at least five virtual face-to-face (video) interactions and at least 10 other interactions either via phone call, email, or text messaging over the 6-month time period.

SUMMARY:
The purpose of this study is to test a peer support intervention for caregivers who are caring for a loved one living with dementia.

DETAILED DESCRIPTION:
African Americans are twice as likely to develop Alzheimer's disease or a related form of dementia (ADRD) than their White counterparts. These individuals are, however, more often diagnosed later, creating additional physical, spiritual, psychosocial challenges for both the person living with ADRD and their family caregivers. African American ADRD caregivers are therefore at greater risk for adverse physiological and psychological health effects of caregiving, including significant burden and stress. Evidence suggests that peer to peer support using storytelling may be effective in assisting ADRD caregivers with surrogate healthcare decision making, an important aspect of palliative care. Access to and use of palliative care, a recognized approach to serious illness care symptom management, among African Americans are low. The impact of this healthcare inequity further reduces the quality of life for African American ADRD caregivers and subsequently their care recipients. Prior approaches to serious illness care have failed to address the needs of African Americans living with ADRD from a palliative care perspective. This inability to meet their needs leads to increased unmet caregiver needs. Peer mentorship, a relationship-centered person-to-person approach may reduce healthcare decision making burden within cultural groups such as African Americans through cultural tailoring by promoting oral traditions, personal contact, and storytelling. Our current study includes perspectives of lower socioeconomic status African American ADRD caregivers who have expressed the need for person-centered, non-judgmental, on-demand, culturally congruent caregiving support for advance care planning and healthcare decision making. Simultaneously, former caregivers retrospectively described perceived benefits of peer support while caregiving and their willingness to serve as peer mentors to current caregivers. Additional data from healthcare provider and community stakeholders support the need and potential benefits of peer support for ADRD caregivers. Based on these preliminary findings, there is an urgent need and exciting opportunity to address the unmet palliative care needs of current caregivers through peer support. For this innovative project, investigators will use the experiential expertise of former caregivers to help current caregivers with advance care planning and healthcare decision making. The purpose of this project is to use a stakeholder-informed approach in further developing and pilot testing the co-created Peer Support for Caregivers of African Americans Living with Alzheimer's Disease and Related Dementias (Pair2Care), a culturally sensitive caregiver peer support intervention.

Aim: Conduct feasibility and acceptability testing of Pair 2 Care in current and trained former African American ADRD family caregiver peers paired based on congruent identity traits (e.g., relationship to care recipient, gender identity, etc.). Investigators will determine if Pair2Care is feasible and acceptable by evaluating satisfaction and appropriateness of the intervention for broader dissemination.

ELIGIBILITY:
Inclusion Criteria:

* African-American
* English-speaking
* Adult (18+)
* Family caregivers of people living with dementia (current or former)

Exclusion Criteria:

* Non-African-American
* Non-English-speaking
* Under age 18
* Non-Family caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University College of Nursing, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moss KO, Tan A, Brody AA, Bullock K, Wright KD, Johnson K, Happ MB. A Peer Support Intervention for Black Family Caregivers of Persons Living With Dementia: A Feasibility Study. J Am Geriatr Soc. 2025 Dec 16. doi: 10.1111/jgs.70241. Online ahead of print. PMID 41403114

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peer Support
Started | 15
Completed | 14
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Peer Support
Number analyzed (Participants) | 15
Age, Customized [Mean (Standard Deviation); unit: years] | 59.6 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Marital Status [Count of Participants; unit: Participants]
  Single | 3
  Separated/Divorced | 3
  Married | 8
  Widowed | 1
Employment [Count of Participants; unit: Participants]
  Full-time | 7
  Part-time | 2
  Homemaker | 1
  Not employed, retired | 5
Relationship to loved one with dementia [Count of Participants; unit: Participants]
  Spouse | 2
  Daughter | 10
  Son | 0
  Other relative | 0
  Friend/Neighbor | 0
  Other | 3
Years as caregiver to the loved one with dementia [Mean (Standard Deviation); unit: years] | 4.4 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Medical Outcomes Study Social Support Survey (MOS SSS)
Description: This instrument contains 19 items that comprise 4 subscales: Emotional/Informational Support, Tangible Support, Affectionate Support, and Positive Social Interaction. Each item is scored on a 5 point Likert scale of 1 ("none of the time") to 5 ("all the time"), with higher scores indicating more social support. Total and subscale scores are in a range of 1-5 calculated by taking the mean across items.
Time Frame: Baseline and 6 months post baseline
Population: 1 participant was not able to complete the intervention due to the death of their spouse
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer Support
Number analyzed (Participants) | 15
score on a scale
  Emotional/Informational Support at Baseline | 3.75 (1.03)
  Emotional/Informational Support at 6 Months: number analyzed (Participants) | 14
  Emotional/Informational Support at 6 Months | 3.79 (0.99)
  Tangible support at Baseline | 3.68 (1.02)
  Tangible support at 6 months: number analyzed (Participants) | 14
  Tangible support at 6 months | 3.50 (1.29)
  Affectionate support at Baseline | 4.22 (0.67)
  Affectionate support at 6 months: number analyzed (Participants) | 14
  Affectionate support at 6 months | 3.95 (0.90)
  Positive social interaction at Baseline | 4.11 (0.72)
  Positive social interaction at 6 months: number analyzed (Participants) | 14
  Positive social interaction at 6 months | 3.98 (0.83)
  Overall social support at Baseline | 3.88 (0.75)
  Overall social support at 6 months: number analyzed (Participants) | 14
  Overall social support at 6 months | 3.77 (0.83)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the 6 month study period
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Peer Support
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT06064955/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT06064955/ICF_001.pdf